CLINICAL TRIAL: NCT06342258
Title: Effects of Cured Bond On Sealant Retention In The Pediatric Population
Brief Title: COES: Curing Order Effects on Sealants
Acronym: COES
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Catherine Pham, Assistant Professor of Clinical Dentistry, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HS-23-00611
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Dental Sealant; Sealant Retention

STUDY DESIGN:
Intervention Model Description: After baseline examination, a randomized generator, will be used in order to issue which side will bonding agent cured prior to sealant placement. Randomization will be a simple randomization, and will be determined by the provider flipping a coin. Randomization will be performed to ensure graders of sealants will be blinded to which side of bond is cured prior to sealant placement.
  Heads indicates the RIGHT side of mouth WILL be cured prior to sealant placement. The left side of the mouth will have bond and sealant cured together after.
  Tails indicates the LEFT side of the mouth WILL be cured prior to sealant placement. The right side of the mouth will not have bond cured prior to sealant placement.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Heads (Experimental): Heads indicates the RIGHT side of mouth WILL be cured prior to sealant placement. The left side of the mouth will have bond and sealant cured together after.
  Interventions: Drug: Ultradent Ultra Seal XT Plus
- Tails (Experimental): Tails indicates the LEFT side of the mouth WILL be cured prior to sealant placement. The right side of the mouth will not have bond cured prior to sealant placement.
  Interventions: Drug: Ultradent Ultra Seal XT Plus

INTERVENTIONS:
Drug: Ultradent Ultra Seal XT Plus — Each child who has erupted, bilateral permanent molars that qualify for the study and agree to participate will have a side (right or left side) of their mouth randomized for bond that will be cured prior to sealant placement. Daily flossing and oral hygiene instructions will be taught to patients of all study groups. Sealant will be placed using a dental suction isolation system, such as DryShield isolation after prophy cup polish with pumice. No enameloplasty will be conducted.

SUMMARY:
Background: Sealants are a great tool in the prevention of caries in the pediatric population. It has been shown that up to 71% of occlusal decay is preventable after a single sealant application in a fissure, and thus is the standard of care due to difficulty for pediatric patients in hygiene, diet, and overall home care until manual dexterity increases.

Purpose: This prospective randomized case control study aims to look at the longevity of sealants with bonding agent cured prior to sealant placement vs those with uncured bond. The study will be performed by USC graduate pediatric personnel.

Methods: A split mouth prospective randomized control study will be performed on pediatric dental patients at Long Beach Memorial's Children's Dental Health Clinic and USC Pediatric Dental Clinic, placing sealants with cured bond on half of a mouth and sealants with uncured bond on the contralateral half. Intraoral photos will be obtained at the initial visit and recalls to evaluate the overall retention/longevity of the sealant placement. The goal of this study is determine which sealant has higher longevity and to provide recommendations for future pediatric dentists regarding sealant procedures.

DETAILED DESCRIPTION:
The primary objective of this prospective randomized control trial is to test the longevity of pit and fissure resin sealants placed with cured bonding agent compared to resin sealants placed with uncured bonding agent over a 2 year period. Sealants will be evaluated at 6 month recall visits (6 month recall, 12 month recall, 18 month recall and 24 month recall), as determined by comparing time lapse intraoral photos and clinical examinations. Secondary objectives of this study aim to look at caries incidence of sealed permanent molars, by monitoring recurrent caries under sealant placement. Additionaly looking at sealant longevity of pit and fissure sealants of hypomineralized versus non hypomineralized molar, classified using Mathu-Muju Wright Classification, with only mildly hypomineralized molars being utilized for the study.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and ASA II children, aged 5 to 14 years who are patients of CDHC and USC with adequate eruption of permanent first or second molars for placement of sealants
* These teeth will not have previous restorations, interproximal lesions, pathology, or occlusal lesions.
* Behavior of the children should be within a Frankl 3 or 4 category, indicating a "positive" and "Definitely Positive" behavior rating, which would allow for safe and controlled execution of the proposed protocol
* Patient must have contralateral molars in the same arch in which sealants can be placed. For example a child with #30 and #19 present will qualify for the study.

Exclusion Criteria

* Any tooth with previous sealant placement
* Children who are allergic or intolerant to sealant material
* Children who cannot tolerate a dental suction isolation system, such as DryShield isolation
* Children who do not complete a prophy cup polish.
* Children who present with banded or bracketed molars
* Patients or Parents who cannot fully understand an English or Spanish Consent/ Assent form.

Withdrawal Criteria

* Patients can withdraw voluntarily at any time.
* Any tooth which has progression of caries beyond ICCMS Category 3 will be withdrawn from the study. These teeth will be treated with appropriate restorative dental treatment according to the standard of care.
* Any qualifying tooth that subsequently requires a restoration due to trauma will be withdrawn from the study.
* Any patient with an adverse reaction to treatment will be withdrawn. This event will be reported to the IRB.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 217 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sealant Longevity | 2 years
  The primary outcome is measuring sealant longevity with intraoral photos and clinical exams. The outcome will be measured as retention (yes/no) and will be evaluated at 4 time points: 6 months, 12 months, 18 months, and 24 months as compared to initial baseline photos taken at treatment day. Patients/parents will be blinded to treatment status. The evaluation of intraoral photos will be performed by blinded practitioners.

SECONDARY OUTCOMES:
Caries | 2 years
  Secondary objectives of this study aim to look at caries incidence of sealed permanent molars, by monitoring recurrent caries under sealant placement.
Molar hypomineralization | 2 years
  Sealant longevity of pit and fissure sealants of hypomineralized versus non hypomineralized molar, classified using Mathu-Muju Wright Classification, with only mildly hypomineralized molars being utilized for the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Herman Ostrow School of Dentistry of USC, Los Angeles, California, United States